CLINICAL TRIAL: NCT05009524
Title: The Interactive Physical and Cognitive Exercise System (iPACES v3) to Benefit Brain Health in Mild Cognitive Impairment (MCI): A Randomized Clinical Trial of Neuro-exergaming Pedal-to-play (iPACES) vs Pedal-while-play (PACE)
Brief Title: The Interactive Physical and Cognitive Exercise System (v3) for Mild Cognitive Impairment (MCI)
Acronym: iPACES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: iPACES LLC (Industry)
Collaborators: Pacific Brain Health Center (Unknown); 1st Playable Productions (Other); Adirondack Neuropsychological Associates (Unknown); Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIA1R44AG071063
Record Dates: First submitted 2021-07-23; First posted 2021-08-17 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: MCI; Mild Cognitive Impairment; Alzheimer Disease; Dementia
Keywords: ADRD; exercise; exergame; physical activity; neuro-exergaming; neuropsychological; cognitive; dual-task; interactive
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Motor Activity | interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: participants are randomly assigned to either iPACES ("pedal-to-play") or PACE ("pedal-while-play") exergaming interventions to be completed 3-5x/wk for 6 months, then PACE crosses over to iPACES and all followed out to 1-year mark
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- iPACES (interactive Physical and Cognitive Exercise System) (Experimental): iPACES (interactive Physical and Cognitive Exercise System) involves a "pedal-to-play" neuro-exergame in which physical and mental exercise are combined in an interactive way. In this condition a person will pedal to control forward motion in a tablet-based game, such as when pedaling along a virtual path and steering to different assigned errand locations.
  Interventions: Device: iPACES (interactive Physical and Cognitive Exercise System)
- PACE (physical and cognitive exercise) (Active Comparator): PACE (Physical and Cognitive Exercise) involves a "pedal-while-play" experience in which physical and mental exercise are combined in a simultaneous, but not fully interactive way. In this condition a person will pedal while also separately steering in a tablet-based game, such as when pedaling while automatically progressing along a virtual path to different assigned errand locations.
  Interventions: Device: PACE (Physical and Cognitive Exercise)

INTERVENTIONS:
Device: iPACES (interactive Physical and Cognitive Exercise System) — iPACES involves a "pedal-to-play" neuro-exergame in which physical and mental exercise are combined in an interactive way. In this condition a person will pedal to control forward motion in a tablet-based game, such as when pedaling along a virtual path and steering to different assigned errand locations.
  Other Names: neuro-exergame
  Arms: iPACES (interactive Physical and Cognitive Exercise System)
Device: PACE (Physical and Cognitive Exercise) — PACE involves a "pedal-while-play" experience in which physical and mental exercise are combined in a simultaneous, but not fully interactive way. In this condition a person will pedal while also separately steering in a tablet-based game, such as when pedaling while automatically progressing along a virtual path to different assigned errand locations.
  Arms: PACE (physical and cognitive exercise)

SUMMARY:
The primary purpose of this study is to attempt to replicate and extend promising pilot findings regarding the cognitive benefits of in-home neuro-exergaming with iPACES (interactive Physical and Cognitive Exercise System v3) for persons with mild cognitive impairment (MCI). Participants will include persons with MCI and their co-residing partner who both exercise at home 3-5 times per week for at least 6 months and are followed through one year. All participation is "remote" (completed at home), with all equipment (pedaler, tablet, etc.) supplied directly to the home, and with all study measures completed via videoconference and mail.

DETAILED DESCRIPTION:
A specific aim is to evaluate the potentially unique contribution of combining mental and physical exercise in an interactive way: "pedal-to-play" (iPACES), as compared with non-interactive, but simultaneous: "pedal-while-play" (PACE).

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of age or older
2. co-residing study partner (spouse, adult child, roommate in same home) willing to participate in the study as an exercising participant as well
3. self or partner meets criteria for MCI (per site staff/MD/neuropsychologist and confirmed by study-administered Montreal Cognitive Assessment; MoCA; score = between 16-26, non-inclusive; Milani, 2018)
4. available for participation for one year (tablet surveys, videoconference evaluations)
5. willing and able to exercise 3-5 times per week for at least 6 months
6. can pedal an under-table elliptical
7. can read off of a small tablet screen
8. proficient in English (speaking and reading for completion of interview, surveys, game)
9. can participate in testing and read and operate tablet touch screen (adequate hearing, vision, speech)
10. written approval from primary care physician and cardiologist (if applicable) to participate in exercise for this study
11. can provide informed consent

Exclusion Criteria:

1. already exercising at recommended levels (45 min of moderate intensity aerobic exercise 5-7x/wk)
2. significant history of cardiovascular problems
3. significant history of stroke
4. significant history of memory problems (e.g., dementia/Alzheimer's)
5. significant history of other neurological condition (e.g., seizures, Parkinson's, etc.)
6. tremor (idiopathic) such that would interfere with touch-screen use required throughout the study (surveys, game-play, etc.)
7. not prone to cybersickness (e.g., "car sickness" or problems with "screen time")
8. cannot provide informed consent (i.e., when phone screened with the Impaired Decision Making Capacity screen)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
executive function | change from baseline to 6 months
  cognitive function composite score from neuropsychological tests (e.g., Stroop)
everyday function | change from baseline to 6 months
  subjective cognitive function in everyday living (e.g., Ecological Validity Scale)

SECONDARY OUTCOMES:
biomarker | change from baseline to 6 months
  biomarker (dried blood spot samples; DBSS) linking exercise to cognitive function (e.g., Brain Derived Neurotrophic Factor)

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — iPACES LLC
Locations (1):
- remote trial conducted via video-conference/mail in-home all locations in the continental USA, Clifton Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be made available in downloadable form
Supporting Information: Study Protocol, CSR
Time Frame: 1-3 years depending upon pace of enrollment
Access Criteria: IPD sharing access may be requested at support@myipaces.org

REFERENCES:
- [Result] Wall K, Stark J, Schillaci A, Saulnier ET, McLaren E, Striegnitz K, Cohen BD, Arciero PJ, Kramer AF, Anderson-Hanley C. The Enhanced Interactive Physical and Cognitive Exercise System (iPACESTM v2.0): Pilot Clinical Trial of an In-Home iPad-Based Neuro-Exergame for Mild Cognitive Impairment (MCI). J Clin Med. 2018 Aug 30;7(9):249. doi: 10.3390/jcm7090249. PMID 30200183
- [Result] Anderson-Hanley C, Stark J, Wall KM, VanBrakle M, Michel M, Maloney M, Barcelos N, Striegnitz K, Cohen BD, Kramer AF. The interactive Physical and Cognitive Exercise System (iPACES): effects of a 3-month in-home pilot clinical trial for mild cognitive impairment and caregivers. Clin Interv Aging. 2018 Sep 4;13:1565-1577. doi: 10.2147/CIA.S160756. eCollection 2018. PMID 30233154
- [Result] Anderson-Hanley C, Barcelos NM, Zimmerman EA, Gillen RW, Dunnam M, Cohen BD, Yerokhin V, Miller KE, Hayes DJ, Arciero PJ, Maloney M, Kramer AF. The Aerobic and Cognitive Exercise Study (ACES) for Community-Dwelling Older Adults With or At-Risk for Mild Cognitive Impairment (MCI): Neuropsychological, Neurobiological and Neuroimaging Outcomes of a Randomized Clinical Trial. Front Aging Neurosci. 2018 May 4;10:76. doi: 10.3389/fnagi.2018.00076. eCollection 2018. PMID 29780318
- [Result] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206
- [Result] Anderson-Hanley C, Maloney M, Barcelos N, Striegnitz K, Kramer A. Neuropsychological Benefits of Neuro-Exergaming for Older Adults: A Pilot Study of an Interactive Physical and Cognitive Exercise System (iPACES). J Aging Phys Act. 2017 Jan;25(1):73-83. doi: 10.1123/japa.2015-0261. Epub 2016 Aug 24. PMID 27337738